CLINICAL TRIAL: NCT03086603
Title: Prospective Observational Study About Variation of Principal Hemodynamic Parameters, Collected With Non-invasive Monitoring, in Patients Undergoing Spinal Anesthesia for Primary Elective Hip Arthroplasty.
Brief Title: Observation of Principal Hemodynamic Variables After Spinal Anesthesia With Non Invasive Hemodynamic Monitoring
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Daniela Ghisi, principal investigator, Istituto Ortopedico Rizzoli
Other Study IDs: EmoSpin
Record Dates: First submitted 2017-02-28; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Hemodynamics; Fluid Therapy; Anesthesia, Spinal; Monitoring, Intraoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is aimed at observe how spinal anesthesia modifies the hemodynamic state of the patient after optimization to preload independence with a Goal Directed Therapy algorithm guided by non invasive hemodynamic monitoring with Clearsight.

DETAILED DESCRIPTION:
This is an observational prospective single group study.

Patients will be monitored with ECG (III leads), non invasive blood pressure cuff (NIBP) cuff, pulse oximetry and Clearsight finger cuff after their arrival in the operating room. Basal Stroke Volume (SV) and indexed Stroke Volume (SVI) will be registered.

The basal value will be optimized according to the study goal directed fluid therapy algorithm: a 200ml fluid challenge will be administered until the SV will increase of at least 10%. When the SV will stop increasing significantly after crystalloid administration, the SV and SVI value will be registered as SVoptimized (SVopt) and SVI optimized (SVIopt), while the same values trigger of the last fluid challenge will be registered as SVtarget1 and SVItarget1. A constant infusion of crystalloids 2 ml/Kg/h will be maintained throughout the study period.

Then, spinal anesthesia will be administered (levobupivacaine 0.5% 0.25mg/kg of ideal weight) in lateral decubitus. After 15 minutes, patients will be turned supine and after 5 minutes SV and SVI will be registered and compared with values SVtarget1 and SVItarget1: if within 10% of range, data will be registered as SVtarget2 and SVItarget2 and patient will maintain basal crystalloid infusion. Otherwise, patients will receive a fluid optimization similar to what described previously before spinal, until values will be within 10% of range of SV and SVI.

Afterwards patients will be transferred to the operating room and will be followed as described in Figure 2. At the end of surgery, patients will be transferred to the Recovery Room and will be monitored and optimized.

When patients will reach an Aldrete's Score ≥ 9/10 and a Bromage's score = 0 with sensibility restored at S1, we will compare SV and SVI value with SVtarget1 and SVItarget1 and treated accordingly.

Spontaneous micturition will be tested and in case a bladder volume > 600ml will be detected with ultrasound before recovery room discharge criteria fulfillment, we will proceed with urinary catheterization.

At patient discharge from the Recovery Room the study will be completed.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective primary hip arthroplasty
* scheduled for spinal anesthesia
* American Society of Anaesthesiologists' (ASA) score 2 or 3
* aged between 50 and 80 years

Exclusion Criteria:

* contraindications to neuraxial anaesthesia
* peripheral vascular abnormalities
* American Society of Anaesthesiologists' (ASA) score 1, 4 and 5
* patients' refusal

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients aged between 50 and 80 years, with an American Society of Anaesthesiologists' (ASA) score 2 or 3 and scheduled for elective primary total hip arthroplasty under spinal anaesthesia. Exclusion criteria were contraindications to neuraxial anaesthesia, peripheral vascular abnormalities (severe vascular diseases, Raynaud's disease, arteriovenous fistula for hemodialysis, previous vascular surgery of the upper arms, advanced diabetes with neuropathy or vascular disease), ASA classes 1, 4 and 5 and patients' refusal.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
stroke volume and stroke volume index | duration of spinal anesthesia procedure
  stroke volume and stroke volume index variation after spinal anesthesia

SECONDARY OUTCOMES:
cardiac output and cardiac index | duration of spinal anesthesia procedure
  cardiac output and cardiac index variation after spinal anesthesia
peripheral vascular resistance index (SVRI) | duration of spinal anesthesia procedure
  peripheral vascular resistance index variation after spinal anesthesia
episodes of hypotension and hypertension intraoperatively | duration of surgery
  variation of Mean Arterial Pressure (MAP) +/- 30% os basal value

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonarelli, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No